CLINICAL TRIAL: NCT00550524
Title: Phase 1 Study of Bone Marrow - Derived Stem Cell for the Treatment of Knee Osteoarthritis
Brief Title: Stem Cell Transplantation for the Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Fereydoun Davatchi, Head Rheumatology Research Center, Rheumatology Research Center, Tehran University for Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3087
Record Dates: First submitted 2007-10-27; First posted 2007-10-30 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Knee osteoarthritis
  Interventions: Biological: Autologous Stem Cell Transplantation

INTERVENTIONS:
Biological: Autologous Stem Cell Transplantation — Autologous bone marrow aspiration (20 ml) from iliac crest. Separation of mononuclear cells using ficoll hypaque and culture in 10% fetal bovine serum and Dulbecco modified eagles medium. After confluent stage, detachment of cells with trypsin/EDTA, and subculture. Repeated passages until obtainment of required cell number. Confluent cells of last passage are washed with tyrode solution and incubate with M199 for 60 minutes. Cells are separated using trypsin/EDTA and washed 3 times with M199 and 1% HSA. Precipitate will be diluted with heparinized M199 to make solution with 6×106 cells /ml. Sample will be tested for viability and detection of CD45, CD34, CD90, CD44, CD13, CD105, and CD166 before injection. The number of cells for injection will be between 20-25 million cells; in a maximum volume of 4-6 ml. Cells will be injected in the knee joint with a 21 gauge needle.

SUMMARY:
The purpose of this study is to find if autologous stem cell transplantation can improve clinical manifestations of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Moderate bilateral knee osteoarthritis

Exclusion Criteria:

* No infectious or inflammatory arthritis

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
1- Comparison of pain in the injected knee with the controlateral knee 2- Comparison of joint motion of the injected knee with the controlateral knee | 12 months

SECONDARY OUTCOMES:
Evaluation of side-effects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fereydoun Davatchi, MD, Study Chair — Rheumatology Research Center, Medical Sciences/University of Teheran; Behrouz Nikbin, MD, Principal Investigator — Department of Immunology, Medical Sciences/University of Tehran
Locations (1):
- Rheumatology Research Center, Behcet's Disease Unit (Shariati Hospital), Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Le Blanc K. [Mesenchymal stem cells. Basic science and future clinical use]. Lakartidningen. 2002 Mar 21;99(12):1318-21, 1324. Swedish. PMID 11998164
- [Background] Caplan AI. Mesenchymal stem cells. J Orthop Res. 1991 Sep;9(5):641-50. doi: 10.1002/jor.1100090504. PMID 1870029
- [Background] Caplan AI, Elyaderani M, Mochizuki Y, Wakitani S, Goldberg VM. Principles of cartilage repair and regeneration. Clin Orthop Relat Res. 1997 Sep;(342):254-69. PMID 9308548
- [Background] Solchaga LA, Welter JF, Lennon DP, Caplan AI. Generation of pluripotent stem cells and their differentiation to the chondrocytic phenotype. Methods Mol Med. 2004;100:53-68. doi: 10.1385/1-59259-810-2:053. PMID 15280587
- [Background] Caplan AI. Adult mesenchymal stem cells for tissue engineering versus regenerative medicine. J Cell Physiol. 2007 Nov;213(2):341-7. doi: 10.1002/jcp.21200. PMID 17620285
- [Derived] Davatchi F, Abdollahi BS, Mohyeddin M, Shahram F, Nikbin B. Mesenchymal stem cell therapy for knee osteoarthritis. Preliminary report of four patients. Int J Rheum Dis. 2011 May;14(2):211-5. doi: 10.1111/j.1756-185X.2011.01599.x. Epub 2011 Mar 4. PMID 21518322